CLINICAL TRIAL: NCT00594152
Title: Anti-Nephropathic Effects of Chronic Intermittent Intravenous Insulin Therapy (CIIIT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: John D'Elia, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS#92-16
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Diabetic Nephropathy; Diabetic Retinopathy
Keywords: Diabetic autonomic neuropathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetic Retinopathy; Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1Control (No Intervention): Standard treatment of type 1 diabetes mellitus with 3-4 subcutaneous injections of insulin daily
- Treatment (Experimental): Intervention: three one-hour courses of pulsed intravenous insulin infusion on a single day per week in addition to standard subcutaneous insulin.
  Interventions: Drug: CIIIT

INTERVENTIONS:
Drug: CIIIT — The intravenous infusion group received three one-hour courses of pulsed intravenous insulin infusion on a single day per week in addition to subcutaneous insulin.
  Arms: Treatment

SUMMARY:
Investigators with the goal of optimizing glycemic and blood pressure control saw type 1 diabetic patients weekly. A control group received 3-4 subcutaneous insulin injections per day; an intravenous insulin pulsed infusion group received, in addition, three one hour infusions in a pulsatile fashion over one eight hour period each week. Patients were followed for 12 months with periodic testing of renal function by repeated blood and urinary analyses; diabetes control by blood testing and diabetes impact measurement score; cardiac and autonomic function by echocardiography, 24 hour electrocardiographic testing; and visual changes with repeated fundus photography. The study hypothesis was that correction of respiratory quotient would correct the defect leading to microvascular complications of diabetes (Type 1).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetics with proteinuria willing to be seen weekly for the evaluation of renal function

Exclusion Criteria:

* Associated active medical diseases that would not permit evaluation of stable renal disease over 18 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 1993-01; Study Completion 1995-01 (Actual)

PRIMARY OUTCOMES:
Rate of loss of creatinine clearance | 18 months

SECONDARY OUTCOMES:
Quality of life assessment | 12 to 18 months
Change in cardiac autonomic function | 12 to18 months
Change in retinal photos | 12 to 18 months
Change in cardiac function | 12 to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: John A D'Elia, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Dailey GE, Boden GH, Creech RH, Johnson DG, Gleason RE, Kennedy FP, Weinrauch LA, Weir M, D'Elia JA. Effects of pulsatile intravenous insulin therapy on the progression of diabetic nephropathy. Metabolism. 2000 Nov;49(11):1491-5. doi: 10.1053/meta.2000.17700. PMID 11092517
- [Derived] Weinrauch LA, Sun J, Gleason RE, Boden GH, Creech RH, Dailey G, Kennedy FP, Weir MR, D'Elia JA. Pulsatile intermittent intravenous insulin therapy for attenuation of retinopathy and nephropathy in type 1 diabetes mellitus. Metabolism. 2010 Oct;59(10):1429-34. doi: 10.1016/j.metabol.2010.01.004. Epub 2010 Mar 1. PMID 20189608